CLINICAL TRIAL: NCT02400723
Title: Reducing Anxiety and Improving Functioning in Older Veterans
Brief Title: Anxiety in Older Veterans
Acronym: BREATHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1478-W; 1IK2RX001478-01A2 (NIH)
Record Dates: First submitted 2015-02-26; First posted 2015-03-27 (Estimated); Results first posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-05

CONDITIONS: Anxiety Disorders
Keywords: behavioral intervention; relaxation; Veterans; geriatric
MeSH Terms: conditions — Anxiety Disorders | interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BREATHE (Experimental): Four weeks of DVD-delivered behavioral intervention. Intervention consists of diaphragmatic breathing and progressive muscle relaxation.
  Interventions: Behavioral: Progressive Muscle Relaxation; Behavioral: Diaphragmatic Breathing
- Psychoeducation (Placebo Comparator): Four weeks of DVD-delivered psychoeducation as an attention placebo control.
  Interventions: Other: Psychoeducation (Placebo)

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation — Progressive Muscle Relaxation is a treatment in which individuals tense and release their muscle groups in a sequential order. This helps reduce anxiety and tension. It also teaches individuals to differentiate between muscle tension and relaxation.
  Other Names: Progressive Relaxation Training
  Arms: BREATHE
Behavioral: Diaphragmatic Breathing — Diaphragmatic breathing is a way in which people breathe using their diaphragm. This type of breathing has been found to promote relaxation and reduce stress.
  Other Names: Deep breathing
  Arms: BREATHE
Other: Psychoeducation (Placebo) — DVD-delivered psychoeducation. Participants will view videos that contain information about what anxiety is and information about one's well-being. This condition is an attention placebo control.
  Arms: Psychoeducation

SUMMARY:
Anxiety leads to poor quality of life, avoidance of activities, decreased social engagement, functional decline, and disability in older patients. This study will compare two self-directed treatments delivered via Digital Versatile Disc (DVD) videos that can be viewed in one's own home. The two treatments being compared are: psychoeducation, which refers to information and education about anxiety, and a behavioral treatment program, called BREATHE (Breathing, Relaxation and Education for Anxiety Treatment in the Home Environment). BREATHE teaches diaphragmatic breathing and progressive muscle relaxation. Participants will be randomly assigned to either treatment. The study is 12 weeks long. There are 4 weeks of treatment via DVD and 8 weeks of follow-up. Participants will be asked questions about anxiety symptoms, mood, health and functioning.

DETAILED DESCRIPTION:
Anxiety is pervasive, costly, and leads to behavioral avoidance, disability, and poor quality of life. The proposed Career Development Award level-2 (CDA-2) study will examine the efficacy of a brief psychosocial intervention for anxiety in older Veterans with anxiety disorders. The psychosocial intervention is called BREATHE (Breathing, Relaxation and Education for Anxiety Treatment in the Home Environment) and teaches diaphragmatic breathing and progressive muscle relaxation via DVD videos that can be viewed in Veterans' own homes. The BREATHE treatment includes age-appropriate vignettes of anxiety-evoking situations. This project is aligned with older adults' preference of psychotherapy to pharmacotherapy for treating anxiety. BREATHE is expected to benefit older Veterans ( 60 years) by reducing anxiety and avoidance and thereby increasing their engagement in activities and improving overall functioning. This aim will be tested in a randomized control trial of DVD-based BREATHE compared with DVD-based psychoeducation in 60 older Veterans with anxiety disorders (Generalized Anxiety Disorder, Panic Disorder, Agoraphobia, Social Anxiety Disorder, and unspecified/other specified anxiety disorder). The study is 12 weeks long with both treatments lasting 4 weeks followed by an 8 week follow-up period. It is hypothesized that BREATHE will result in a statistically and clinically significant reduction of anxiety symptoms as measured with the Geriatric Anxiety Scale compared with psychoeducation. Improvements in functioning (Activity Card Sort) are expected for participants randomized to the BREATHE condition compared with those randomized to psychoeducation. Hypotheses in will be addressed with mixed effects models.

ELIGIBILITY:
Inclusion Criteria:

* Veterans aged 60 years or older.
* Meets criteria for an anxiety disorder (Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia, Anxiety Disorder Unspecified, Anxiety Disorder Other Specified).
* English-speaking.

Exclusion Criteria:

* Diagnosis of dementia or significant cognitive impairment as determined by a brief cognitive screen.
* Diagnosis of serious mental illness (bipolar disorder, psychosis, schizophrenia),
* taking benzodiazepines more than once a week per self report.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Gould, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gould CE, Carlson C, Wetherell JL, Goldstein MK, Anker L, Beaudreau SA. Brief Video-Delivered Intervention to Reduce Anxiety and Improve Functioning in Older Veterans: Pilot Randomized Controlled Trial. JMIR Aging. 2024 Dec 9;7:e56959. doi: 10.2196/56959. PMID 39652863

RESULTS

PARTICIPANT FLOW:
Groups:
- BREATHE: Four weeks of video-delivered behavioral intervention. Intervention consists of diaphragmatic breathing and progressive muscle relaxation.
  Progressive Muscle Relaxation: Progressive Muscle Relaxation is a treatment in which individuals tense and release their muscle groups in a sequential order. This helps reduce anxiety and tension. It also teaches individuals to differentiate between muscle tension and relaxation.
  Diaphragmatic Breathing: Diaphragmatic breathing is a way in which people breathe using their diaphragm. This type of breathing has been found to promote relaxation and reduce stress.
- Psychoeducation: Four weeks of video-delivered psychoeducation as an attention placebo control.
  Psychoeducation (Placebo): video-delivered psychoeducation. Participants will view videos that contain information about what anxiety is and information about one's well-being. This condition is an attention placebo control.
Period: Overall Study
Arm/Group | BREATHE | Psychoeducation
Started | 27 | 29
Completed | 22 | 24
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BREATHE | Psychoeducation | Total
Number analyzed (Participants) | 27 | 29 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 7 | 10
  >=65 years | 24 | 22 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.8 (6.2) | 70.0 (6.0) | 71.4 (6.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 23 | 25 | 48
  Female | 3 | 4 | 7
  Unknown | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 22 | 21 | 43
  Unknown or Not Reported | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 18 | 21 | 39
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 29 | 56
Geriatric Anxiety Scale [Mean (Standard Deviation); unit: units on a scale] — The Geriatric Anxiety Scale (GAS) is a 30-item measure of somatic, cognitive, and affective symptoms of anxiety. The first 25 items of the measure are used to compute the total score; the last 5 items provide information about the content of worries or fears. Participants provide severity ratings for items using on a four-point Likert-type scale. Scores range from 0 to 75; higher scores indicate more severe anxiety.
  units on a scale | 17.1 (10.4) | 18.8 (10.5) | 18.0 (10.4)
Patients Health Questionnaire 9-item [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire 9-item (PHQ-9) is a 9-item depression assessment rated on a four-point Likert-type scale with scores ranging from 0 to 27. Higher scores indicate more severe depression. It includes one item that inquires about suicide ideation. Validity and reliability have been established with primary care patients.
  units on a scale | 7.4 (6.1) | 6.7 (4.6) | 7.0 (5.3)
Hamilton Anxiety Scale [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Anxiety Scale (HAM-A) a clinician-administered rating scale, assesses the severity of anxiety using 14-items rated on a five-point scale ranging from 0 to 4. Scores range from 0 to 56 with higher scores indicative of more severe anxiety.
  units on a scale | 18.0 (7.6) | 16.6 (7.1) | 17.3 (7.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Anxiety Symptoms
Description: The Geriatric Anxiety Scale (GAS) (Segal et al., 2010) is a 30-item measure of somatic, cognitive, and affective symptoms of anxiety. The first 25 items of the measure are used to compute the total score; the last 5 items provide information about the content of worries or fears. Participants provide severity ratings for items using on a four-point Likert-type scale. Scores range from 0 to 75; higher scores indicate more severe anxiety.
Time Frame: Change from baseline at 12 weeks
Population: Discrepancy is due to some participants missing post-assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE | Psychoeducation
Number analyzed (Participants) | 22 | 24
units on a scale | 1.77 (9.29) | -2.42 (7.88)

2. Primary Outcome: Change in Activity Engagement
Description: The Activity Card Sort (ACS; Baum & Edwards, 2001) contains 80 photographs that depict the performance of instrumental activities, low-physical-demand leisure activities, high-physical-demand leisure activities, and social activities. This measure will be used to assess engagement in activities. A lifestyle adjusted performance score was calculated on this measure. Scores show of the total activities ever performed in one's life, what percentage are currently performed (0% to 100%). Lower percentages would suggest that individuals are no longer performing activities that they used to do.
Time Frame: Change from baseline at 12 weeks
Population: Following the onset of the coronavirus pandemic, the research team switched to virtual administration of pre and post measurements with institutional review board approval. This measure was unable to be obtained during these virtual assessments as it required a card sorting procedure that could not be completed by telephone (n = 15 assessments missing due to COVID, n = 1 did not complete measure at baseline; n = 7 missing post assessments including this measure)
Measure: Mean (Standard Deviation); unit: percentage of activities
Arm/Group | BREATHE | Psychoeducation
Number analyzed (Participants) | 15 | 18
percentage of activities | 2.74 (8.71) | .71 (10.42)

3. Primary Outcome: Change in Anxiety Symptoms
Description: The Geriatric Anxiety Scale (GAS) (Segal et al., 2010) is a 30-item measure of somatic, cognitive, and affective symptoms of anxiety. The first 25 items of the measure are used to compute the total score; the last 5 items provide information about the content of worries or fears. Participants provide severity ratings for items using on a four-point Likert-type scale. Scores range from 0 to 75; higher scores indicate more severe anxiety. This outcome will be used to examine the effects of the 4 week BREATHE treatment.
Time Frame: Change from baseline at 4 weeks
Population: Five participants in the BREATHE group were missing week 4 assessments; 1 participant in Psychoeducation was missing a week 4 assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE | Psychoeducation
Number analyzed (Participants) | 22 | 28
units on a scale | 1.45 (6.40) | -4.75 (9.72)

4. Secondary Outcome: Change in Clinician-rated Anxiety Symptoms
Description: The Hamilton Anxiety Scale (HAM-A), a clinician-administered rating scale, assesses the severity of anxiety using 14-items rated on a five-point scale ranging from 0 to 4. It has adequate internal consistency, high inter-rater reliability, and good-to-adequate concurrent validity. The Structured Interview Guide for Hamilton Anxiety Scale provides descriptive anchors to guide clinician decision making ratings based on both frequency and severity. Scores range from 0 to 56 with higher scores indicative of more severe anxiety.
Time Frame: Change from baseline at 12 weeks
Population: Eight participants were missing post-assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE | Psychoeducation
Number analyzed (Participants) | 22 | 24
units on a scale | -2.36 (6.36) | -.042 (7.10)

5. Secondary Outcome: Change in Functioning
Description: The Veterans Research and Development Corporation (RAND) 12-Item Health Survey (VR-12) is a 12-item measure that assesses mental and physical health and functioning. It is validated for use with Veterans. The measure includes subjective ratings of one's health and assessments of functioning for the past four weeks. We used the mental health functioning component of the VR-12. The VR-12 scores are standardized using a T-score metric with a mean of 50 and a standard deviation of 10. Scores range from 0 (worst possible outcome) to 100 (best possible outcome).
Time Frame: Change from baseline at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE | Psychoeducation
Number analyzed (Participants) | 22 | 24
units on a scale | -.09 (2.45) | -.67 (2.73)

6. Other Pre Specified Outcome: Change in Anxiety Control
Description: The Anxiety Control Questionnaire (ACQ) (Rapee et al., 1996) is a 30-item self-report measure assessing one's perceived ability to control anxiety-evoking situations and emotional reactions to these situations. Each item is scored using a Likert-type scale with values ranging from 0 (strongly disagree) to 5 (strongly agree). Total scores range from 0 to 150. Higher scores indicate greater perceived control over one's anxiety. This measure assess aspects of avoidance and was included to examine whether BREATHE has an effect on perceived anxiety control compared with the psychoeducation control condition. This questionnaire asks participants to indicate how typical each statement is of themselves.
Time Frame: Change from baseline at 12 weeks
Population: 8 participants were missing post assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE | Psychoeducation
Number analyzed (Participants) | 23 | 25
units on a scale | 6.35 (24.86) | 5.76 (20.06)

7. Other Pre Specified Outcome: Change in Depressive Symptoms
Description: The Patient Health Questionnaire 9-item (PHQ-9) is a 9-item depression assessment rated on a four-point Likert-type scale with scores ranging from 0 to 27. Higher scores indicate more severe depression. It includes one item that inquires about suicide ideation. Validity and reliability have been established with primary care patients.
Time Frame: Change from baseline at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE | Psychoeducation
Number analyzed (Participants) | 22 | 24
units on a scale | .00 (4.08) | -.21 (3.09)

8. Other Pre Specified Outcome: Comorbidity
Description: The Cumulative Illness Rating Scale for Geriatrics (CIRS-G) was selected to measure comorbidity. The CIRS-G assesses severity of conditions important to older adults' functional status and well-being, such as arthritis, that are impairing yet not fatal. Raters will examine the severity of 14 medical problem categories. Categories include the severity of present illness and the consideration of past medical history. Each of 14 categories are rated on a scale from 0 to 4. Total scores range from 0 to 56 with higher scores. The severity scores reported here represent the total score divided by the total number of categories endorsed. Higher scores indicate more severe illness. This construct of comorbidity is being examined as a potential moderator of treatment outcomes in exploratory analyses.
Time Frame: Baseline
Population: 55 of 56 participants gave permission to review their medical records to derive this rating.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE | Psychoeducation
Number analyzed (Participants) | 26 | 29
units on a scale | 1.59 (.29) | 1.57 (.30)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | BREATHE | Psychoeducation
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/29
Other Adverse Events (participants affected / at risk) | 1/27 | 0/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BREATHE (N=27) | Psychoeducation (N=29)
Abdominal pain, muscle strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Strained muscle in abdomen, stomach discomfort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT02400723/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT02400723/ICF_001.pdf